CLINICAL TRIAL: NCT06776406
Title: Real-Time Head Stabilization of Patients Undergoing Radiation Therapy
Brief Title: Head Stabilization in Whole Brain RT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant ended
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02323; 855442 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2024-09-04; First posted 2025-01-15 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Brain Cancer
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Head Stabilization (Experimental): Real-time patient head stabilization during radiation therapy will be performed using a specially designed patient mask and head holder that are connected to a robotic patient support platform (Freedom Pursuit Robotic Platform, CDR Systems, Canada) that will use real-time 3D surface data from the AlignRT system (3D surface imager) as an input and will perform small sub-millimeter corrections.
  Interventions: Device: Freedom Pursuit Robotic Platform

INTERVENTIONS:
Device: Freedom Pursuit Robotic Platform — The Freedom Pursuit Robotic Platform is a robotic head holder device that uses data from the AlignRT system (3D surface imager) to make small movements of a patient's head to stabilize it during radiation therapy.

SUMMARY:
This is a single-center, single-arm observational study in which the investigators aim to develop an advanced motion control system for head stabilization in patients undergoing whole brain radiation therapy.

DETAILED DESCRIPTION:
Standard of care treatment is to be immobilized with a mask for whole brain radiation therapy. The purpose of this study is to develop a process to track and correct a person's head movements in real time during radiation treatment. To do this, the investigators will use a mask and head holder connected to a robotic support platform which can make small movements of the head holder.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and older undergoing whole brain radiation therapy
* Participants must sign the informed consent form

Exclusion Criteria:

All patients not meeting the above inclusion criteria will not be considered for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-14 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2025-10-14 (Actual)

PRIMARY OUTCOMES:
Robotic Head Holder Stabilization During Radiation Therapy | 24 months
  The total percentage of time that a participant is positioned ≤ 0.5mm and ≤ 0.5deg within target during radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Alonso-Basanta, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No